CLINICAL TRIAL: NCT01017653
Title: Phase II Study of Panitumumab in Combination With Irinotecan for Malignant Gliomas
Brief Title: Panitumumab and Irinotecan for Malignant Gliomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study did not reach benchmark efficacy rule at 16 subjects
Sponsor: Annick Desjardins (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Assist Professor of Medicine-Neurology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00015447
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-07

CONDITIONS: Malignant Glioma of Brain
Keywords: Panitumumab; Vectibix; Irinotecan; CPT-11; Camptosar; Malignant glioma; Glioblastoma multiforme; Gliosarcoma; Duke; Vredenburgh; Pro00015447
MeSH Terms: conditions — Glioma; Glioblastoma; Gliosarcoma | interventions — Irinotecan; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab and irinotecan (Experimental)
  Interventions: Drug: Irinotecan; Drug: Panitumumab

INTERVENTIONS:
Drug: Irinotecan — Irinotecan: for those patients on an enzyme-inducing anti-epileptic drug (EIAED), irinotecan will be dosed at 340 mg/m2 every other week. For those not on an EIAED, irinotecan will be dosed at 125 mg/m2. Treatment on both drugs will continue until tumor progression or unacceptable toxicity.
  Other Names: Camptosar; CPT-11
Drug: Panitumumab — Panitumumab, 6 mg/kg, as an intravenous infusion every other week. Treatment on both drugs will continue until tumor progression or unacceptable toxicity.
  Other Names: Vectibix

SUMMARY:
This is a phase II study of the combination of panitumumab with irinotecan in malignant glioma patients. The primary objective of the study is to determine the activity of the combination of panitumumab with irinotecan as measured by 6-month progression-free survival. Secondary objectives include the following- to determine the safety of panitumumab in combination with irinotecan in patients with malignant glioma; to determine the effect of panitumumab in combination with irinotecan on corticosteroid dose for each patient; to explore any relationship between epidermal growth factor receptor (EGF-R) mutational analysis and efficacy or toxicity; and, to determine the response rate and overall survival of recurrent glioblastoma (GBM) patients treated with panitumumab in combination with irinotecan.

The patients will have histologically documented grade 4 malignant gliomas (glioblastoma multiforme or gliosarcoma) that have failed at least one prior chemotherapy regimen and all patients will have received radiation therapy. This study will investigate second or greater line of therapy for recurrent grade 4 malignant glioma. The patient population will include 32 patients.

The patients will undergo a baseline magnetic resonance imaging (MRI) as well as a MRI after every six-week cycle to determine response and progression. After 16 patients with recurrent GBM are treated, an interim analysis will be conducted. The most common side effects associated with panitumumab have been dermatological (skin) problems such as erythema (redness of the skin), acneiform rash (skin eruptions of the face), skin exfoliation, pruritus (itching), skin fissures (skin tears), xerosis (dryness of the eye, skin, or mouth), and rash. The most common side effects associated with irinotecan have been decreased blood counts of platelets (increased risk of bleeding), white blood cells (increased risk of infection), red blood cells (anemia); diarrhea, constipation, nausea, vomiting, tiredness, fever, mouth sores, dehydration (excessive loss of body fluids), rash, itching, changes in skin color, swelling, numbness, tingling, dizziness, confusion, low blood pressure, sweating, hot flashes, hair loss, inflammation of the liver, flu-like symptoms, decreased urine output, shortness of breath, and pneumonia (inflammatory disease of the lungs).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of primary malignant glioma (glioblastoma multiforme or gliosarcoma). Patients with recurrent disease whose diagnostic pathology confirmed grade IV malignant glioma (glioblastoma multiforme or gliosarcoma) will not need re-biopsy.
* Age ≥ 18 years.
* Evidence of measurable recurrent or residual primary central nervous system (CNS) neoplasm on contrast-enhanced MRI
* An interval of at least 4 weeks between prior surgical resection, or major surgery requiring general anesthesia or 1 week between prior biopsy or minor surgical procedures and study enrollment. The subjects must have recovered from all surgery related toxicities.
* An interval of at least 12 weeks between prior radiotherapy or 4 weeks from prior monthly chemotherapy, or 7 days from daily chemotherapy.
* The lab values following the prior chemotherapy must return to the baseline prior to study enrollment.
* Karnofsky ≥ 70%.
* Hematocrit ≥ 29%, absolute neutrophil count (ANC) ≥ 1,500 cells/μl, platelets ≥ 125,000 cells/μl.
* Serum creatinine ≤ 1.5 mg/dl, serum magnesium, potassium, calcium, chloride, and sodium ≥ the lower limit of normal, serum glutamic-oxaloacetic transaminase (SGOT) and bilirubin ≤ 1.5 times upper limit of normal.
* Signed informed consent approved by the Institutional Review Board prior to patient entry.
* If sexually active, patients will take contraceptive measures for the duration of the treatments, and for 6 months afterwards.

Exclusion Criteria:

* Pregnancy or breast feeding
* Co-medication that may interfere with study results; e.g. immuno¬suppressive agents other than corticosteroids.
* Active infection requiring intravenous antibiotics.
* uridine diphosphate glucuronosyltransferase 1A1 (UGT1A1) homozygous for the 7/7 genotype.
* Pre-existing diarrhea greater than Grade 1.

Panitumumab-Specific Concerns:

[Subjects meeting any of the following criteria are ineligible for study entry]

* Prior anti-epidermal growth factor receptor (EGFr) antibody therapy or treatment with small molecule EGFr inhibitors
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with the study participation or investigational product(s) administration or may interfere with the interpretation of the results.
* Subject unwilling or unable to comply with study requirements
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, acute or chronic active hepatitis B infection(testing is not required in the absence of clinical suspicion)
* Patients with a history of deep venous thrombosis, pulmonary embolism or on therapeutic anti-coagulation.
* Known allergy or hypersensitivity to any component of the study treatment(s)
* Active infection requiring systemic intravenous treatment of any uncontrolled infections ≤14 days prior to enrollment/randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Groups:
- Panitumumab and Irinotecan: Panitumumab in Combination with Irinotecan : Panitumumab, 6mg/kg, as an intravenous infusion every other week in combination with Irinotecan (dose dependent upon whether the patient is taking an enzyme-inducing anti-epileptic drug [EIAED]). On an enzyme-inducing anti-epileptic drug (EIAED), irinotecan will be dosed at 340 mg/m2 every other week. Not on an EIAED, irinotecan will be dosed at 125 mg/m2. Treatment will continue until tumor progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Panitumumab and Irinotecan
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Panitumumab and Irinotecan
Number analyzed (Participants) | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 48.73 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival (PFS)
Description: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to the Macdonald criteria, or to death due to any cause. Macdonald criteria are standard criteria in neuro-oncology. Tumor assessment was made according to the adapted MacDonald criteria based on the combined evaluation of: 1) assessment of the MRI scan for measurable, evaluable, and new lesions (made by the independent external expert too), 2) overall assessment of neurological performance (made by the investigator), and 3) concomitant steroid use (as reported by the investigator).
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab and Irinotecan
Number analyzed (Participants) | 16
percentage of participants | 12.5 [2.1 to 32.8]

2. Secondary Outcome: One-Year Overall Survival
Description: Percentage of participants surviving 12 months from the start of study treatment. OS was defined as the time from the date of study treatment initiation to the date of the death due to any cause.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab and Irinotecan
Number analyzed (Participants) | 16
percentage of participants | 12.5 [2.1 to 32.8]

3. Secondary Outcome: Safety of Panitumumab in Combination With Irinotecan
Description: Number of participants experiencing a toxicity ≥ grade 3 as graded per CTCAE v.3.0
Time Frame: 16 months
Measure: Number; unit: participants
Arm/Group | Panitumumab and Irinotecan
Number analyzed (Participants) | 16
participants | 10

4. Secondary Outcome: Effect of Panitumumab in Combination With Irinotecan on Corticosteroid Dose
Description: Average change in corticosteroid dose from baseline to the end of cycle 1.
Time Frame: Baseline and Day 29
Population: Insufficient data to analyze the effect of the treatment regimen on corticosteroid dose. Data was not collected for this outcome.
Measure: Number; unit: mg
Arm/Group | Panitumumab and Irinotecan
Number analyzed (Participants) | 16
mg | NA — Insufficient data to analyze the effect of the treatment regimen on corticosteroid dose. Data was not collected for this outcome.

5. Secondary Outcome: Relationship Between Epidermal Growth Factor Receptor (EGF-R) Mutational Analysis and Efficacy or Toxicity
Description: Number of participants with an abnormal fluorescence in situ hybridization (FISH) interpretation that 1) survived < 6 months and 2) experienced a ≥ grade 3 toxicity as graded per CTCAE v.3.0
Time Frame: 16 months
Population: Insufficient data to analyze the relationship between EGF-R analysis and efficacy or toxicity. Data was not collected for this outcome.
Measure: Number; unit: participants
Arm/Group | Panitumumab and Irinotecan
Number analyzed (Participants) | 16
participants
  Abnormal FISH Interpretation & Survived <6 months | NA — Insufficient data to analyze the relationship between EGF-R analysis and efficacy or toxicity
  Abnormal FISH Interpretation & ≥ grade 3 toxicity | NA — Insufficient data to analyze the relationship between EGF-R analysis and efficacy or toxicity

6. Secondary Outcome: Objective Response Rate
Description: Number of participants with an objective response (complete response or partial response) based on modified Macdonald criteria. A complete response is defined as the disappearance of all enhancing rumor and mass effect, off all corticosteroids, accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks. A partial response is defined as greater than or equal to 50% reduction in tumor size on MR (magnetic resonance) / CT(computed tomography) by bi-dimensional measurement on a stable or decreasing dose of corticosteroids, accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks.
Time Frame: 16 months
Population: 2 patients' response was unknown due to withdrawal from the study before an MRI was performed.
Measure: Number; unit: participants
Arm/Group | Panitumumab and Irinotecan
Number analyzed (Participants) | 14
participants | 0

7. Secondary Outcome: Median Overall Survival (OS)
Description: Time in months from the start of study treatment to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab and Irinotecan
Number analyzed (Participants) | 16
months | 4.6 [4.0 to 5.8]

ADVERSE EVENTS:
Time Frame: 16 months
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov
Arm/Group | Panitumumab and Irinotecan
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab and Irinotecan (N=16)
Intracranial hemorrhage (Nervous system disorders) | 1
Ischemia cerebrovascular (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab and Irinotecan (N=16)
"Ear and labyrinth disorders - Other, specify: Pop noise in ears" (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 1
Optic nerve disorder (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
"Gastrointestinal disorders - Other, specify: Acid Reflux" (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 13
Fever (General disorders) | 1
Lung infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 4
Scrotal infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2
"Musculoskeletal and connective tissue disorder - Other, specify: Fall" (Musculoskeletal and connective tissue disorders) | 4
Ataxia (Nervous system disorders) | 3
Cognitive disturbance (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 3
"Nervous system disorders - Other, specify: Concentration impairment" (Nervous system disorders) | 1
"Nervous system disorders - Other, specify: Gait" (Nervous system disorders) | 2
Pyramidal tract syndrome (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 5
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
"Skin and subcutaneous tissue disorders - Other, specify: Cuticle cuts/open wounds" (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders-Other, specify: Increased hair growth (Skin and subcutaneous tissue disorders) | 1
"Skin and subcutaneous tissue disorders - Other, specify: Laceration, head" (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes